CLINICAL TRIAL: NCT03640871
Title: Assessment of Efficacy, Tolerance and Acceptability for the Wound Dressing URGO AWC_019 in the Local Treatment of Acute Wounds, Chronic Wounds and Epidermolysis Bullosa Skin Lesions
Brief Title: HEAL Study: Healing Results, Efficacy and Acceptability of a New Contact Layer
Acronym: HEAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratoires URGO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F-18-06-AWC019
Record Dates: First submitted 2018-08-03; First posted 2018-08-21 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-07

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- URGO AWC_019 dressing (AWC=Advanced Wound Care) (Experimental): URGO AWC_019 dressing (AWC=Advanced Wound Care)
  Interventions: Device: URGO AWC_019 dressing (AWC=Advanced Wound Care)

INTERVENTIONS:
Device: URGO AWC_019 dressing (AWC=Advanced Wound Care) — URGO AWC_019 dressing 10x10 cm (AWC=Advanced Wound Care)

SUMMARY:
Assessment of efficacy, tolerance and acceptability for the wound dressing URGO AWC_019 in the treatment of acute wounds, chronic wounds and epidermolysis bullosa skin lesions

DETAILED DESCRIPTION:
Non-comparative clinical study, conducted in France, to evaluate efficacy, tolerance and acceptability for the wound dressing URGO AWC_019 in the treatment of acute wounds, chronic wounds and epidermolysis bullosa skin lesions

ELIGIBILITY:
Inclusion Criteria:

A. Related to every wounds types:

* Patient over 18 years old who has provided his/her written informed consent
* Patient affiliated to the French Social insurance
* Patient who can be monitored by the same investigation team throughout the whole duration of the study,
* Acute wound (postoperative non-cavitary and non-sutured wound, superficial, middle or deep second degree burn, dermabrasion) or chronic wound (venous or mixed leg ulcer, pressure ulcer) or epidermolysis bullosa skin lesion
* Use of a contact layer as a primary dressing justified by the wound

B. Related to leg ulcer:

* Venous leg ulcer or mixed leg ulcer, i.e. with an Ankle Brachial Pressure Index (ABPI) not less than 0.7 and not more than 1.3, (0.7≤ABPI≤ 1.3)
* Patient who agrees to wear an effective venous compression system every day, associated with the trial dressing

C. Related to pressure ulcer:

* Stage 2, 3 according to the EPUAP (European Pressure Ulcer Advisory Panel) classification system
* Wound on the pelvis (trochanter, ischio or sacrum) or on the heel

Exclusion Criteria:

* Patient under authorship or guardianship
* Woman of child-bearing potential who has no effective contraception method
* Pregnant or breastfeeding woman
* Patient taking part in another clinical trial
* Patient with a known allergy to carboxymethylcellulose (hydrocolloid),
* Patient with a severe illness that might lead to the premature discontinuation of the trial before the 4 weeks of treatment
* Wound requiring surgical treatment or for which surgery is scheduled during the 4 weeks after inclusion
* Patient with an evolving neoplasia condition, treated by radiotherapy, chemotherapy or hormone therapy
* Malignant wound
* Patient with a systemic infection not controlled by suitable antibiotic treatment,
* Wound which is clinically infected

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Relative evolution of the wound surface (in %) at week 4 | 4 weeks
  Relative evolution of the wound surface (in %) at week 4

SECONDARY OUTCOMES:
- Pain on wound URGO AWC_019 dressing removal (measured thanks to Analogical Visual Scale: no pain = 0 mm and unbearable pain = 100 mm) | 4 weeks
  - Pain on wound URGO AWC_019 dressing removal (measured thanks to Analogical Visual Scale: no pain = 0 mm and unbearable pain = 100 mm)
- Wound dressing safety (occurrence of adverse events) | 4 weeks
  - Wound dressing safety (occurrence of adverse events)
- Percentage of healed wounds (healing rate) after 4 weeks of treatment | 4 weeks
  - Percentage of healed wounds (healing rate) after 4 weeks of treatment
- Wound healing time (in days) | 4 weeks
  - Wound healing time (in days)

IPD SHARING:
Plan to Share IPD: No